CLINICAL TRIAL: NCT00358163
Title: Phase I Study of the Oral Vascular Endothelial Growth Factor Inhibitor PTK787/ZK 222584 in Combination With Paclitaxel in Patients With Advanced Solid Tumors.
Brief Title: Trial of PTK787/ZK 222584 Plus Paclitaxel
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Novartis Pharmaceuticals (Industry); Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-046
Record Dates: First submitted 2006-07-28; First posted 2006-07-31 (Estimated); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Metastatic Non-hematologic Malignancies
Keywords: angiogenesis; taxane; tyrosine kinase; pharmacokinetics; Vatalanib; Taxol
MeSH Terms: interventions — vatalanib; Paclitaxel

ARMS (1):
- PTK787/ZK 222584 (Experimental)
  Interventions: Drug: PTK787/ZK 222584; Drug: paclitaxel

INTERVENTIONS:
Drug: PTK787/ZK 222584 — Taken in tablet form daily
  Other Names: Vatalanib
Drug: paclitaxel — Given as a 3-hour infusion once every 21 days

SUMMARY:
PTK787/ZK 222584 is an inhibitor of VEGFR family tyrosine kinases. The primary objective of this study is to assess the safety of daily oral PTK787/ZK 222584 in combination with paclitaxel infused every 21 days. Secondary objectives include pharmacokinetic assessment of the impact of PTK787/ZK 222584 on paclitaxel metabolism and evaluation of tumor response to the investigational treatment.

DETAILED DESCRIPTION:
* We are looking for the highest dose of Paclitaxel that can be given safely in combination with the highest safe dose of Vatalanib. Therefore, not all people will receive the same dose of the study drug.
* Small groups of people will be enrolled in steps on this trial. This first group will be given a certain dose of Paclitaxel and Vatalanib. If they have few or manageable side effects, the next small group of people enrolled will receive higher doses of the study drugs. This increase in doses will continue until the study doctors find the highest dose of the drugs that can be given without causing severe or unmanageable side effects.
* In this study, Vatalanib tablets are taken daily, and paclitaxel is given by three-hour intravenous infusion once every 21 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced solid tumors for whom there is no potentially curative treatment (surgery, radiation therapy or chemotherapy).
* Measurable or non-measurable disease
* Age ≥ 18 years old
* ECOG Performance Status 0 -1
* Laboratory values ≤ 14 days weeks prior to starting study treatment:
* Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L (≥ 1500/mm3)
* Platelets (PLT) ≥ 100 x 109/L (≥ 100,000/mm3)
* Hemoglobin (Hgb) ≥ 9 g/dL
* Serum creatinine ≤ 1.5 ULN
* Serum bilirubin ≤ 1.0 x ULN
* Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) ≤ 2.5 x ULN (≤ CTC grade 1).
* Negative for proteinuria based on dip stick reading OR, if documentation of +1 result for protein on dip stick reading, then total urinary protein ≤ 500 mg and measured creatinine clearance (CrCl) ≥ 50 mL/min from a 24-hour urine collection
* Women of child-bearing age must have a negative serum or urine test.
* Life expectancy ≥ 12 weeks
* Written informed consent obtained
* Resolution of toxicity from previous chemotherapy to ≤ Grade I.
* QTc interval ≤ 0.45 seconds (men) or ≤ 0.47 seconds (women).

Exclusion Criteria:

* Previous hypersensitivity reaction to taxanes or cremophor.
* History or presence of central nervous system (CNS) disease (i.e., primary brain tumor, malignant seizures, CNS metastases or carcinomatous meningitis).
* Prior chemotherapy ≤ 4 weeks prior to registration. Prior nitrosoureas or mitomycin C ≤ 6 weeks prior to registration.
* Prior biologic or immunotherapy ≤ 2 weeks prior to registration. Patients must have recovered from all therapy-related toxicities
* Prior radiotherapy ≤ 4 weeks prior to registration. Patients must have recovered from all therapy-related toxicities. The site of previous radiotherapy should have evidence of progressive disease if this is the only site of disease
* Major surgery (i.e., laparotomy) ≤ 4 weeks prior to registration. Minor surgery ≤ 2 weeks prior to registration. Insertion of a vascular access device is not considered major or minor surgery in this regard. Patients must have recovered from all surgery-related toxicities
* Patients who have received investigational drugs ≤ 4 weeks prior to registration.
* Peripheral neuropathy with functional impairment ≥ CTC grade 2 neuropathy, regardless of causality.
* Pleural effusion or ascites that causes respiratory compromise (≥ CTC grade 2 dyspnea)
* Female patients who are pregnant or breast-feeding, or adults of reproductive potential who are not employing an effective method of birth control. Barrier contraceptives must be used throughout the trial in both sexes. Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are therefore not considered effective for this study. Please refer to appendix for a list of examples of substrates of human liver microsomal P450 enzymes
* Any of the following concurrent severe and/or uncontrolled medical conditions which could compromise participation in the study:
* Uncontrolled high blood pressure, history of labile hypertension, or history of poor compliance with an antihypertensive regimen
* Unstable angina pectoris
* Symptomatic congestive heart failure
* Myocardial infarction ≤ 6 months prior to registration and/or randomization
* Serious uncontrolled cardiac arrhythmia
* Uncontrolled diabetes
* Active or uncontrolled infection
* Interstitial pneumonia or extensive and symptomatic interstitial fibrosis of the lung
* Acute or chronic liver disease (eg., hepatitis, cirrhosis)
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of PTK787/ZK 222584 (i.e., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, bowel obstruction, or inability to swallow the tablets)
* Patients with confirmed diagnosis of human immunodeficiency virus (HIV) infection are excluded at the investigator's discretion if he/she feels that 1) a potential drug interaction between PTK787/ZK 222584, paclitaxel and any of the patient's anti-HIV medications could influence the efficacy of the anti-HIV medication, or 2) it may place the patient at risk due to the pharmacologic activity of PTK787/ZK 222584. Please refer to appendix for a list of examples of substrates of human liver microsomal P450 enzymes
* Patients who are taking therapeutic warfarin sodium (Coumadin) or similar oral anticoagulants that are metabolized by the cytochrome P450 system. Heparin products are allowed. Please refer to appendix for a list of examples of substrates of human liver microsomal P450 enzymes
* Patients unwilling to or unable to comply with the protocol
* Use of recombinant G-CSF products (Neupogen, Neulasta) within three weeks of registration. Chronic use of recombinant erythropoietin is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2006-04-26 (Actual); Primary Completion 2008-05-29 (Actual); Study Completion 2008-05-29 (Actual)

PRIMARY OUTCOMES:
Safety of PTK787/ZK 222584 in combination with paclitaxel | 2 years

SECONDARY OUTCOMES:
Pharmacokinetic effect of PTK787/ZK 222584 on paclitaxel metabolism. Clinical tumor response to study treatment. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Pankaj Bhargava, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts